CLINICAL TRIAL: NCT01268072
Title: A Prospective Observational Study to Evaluate Biomarkers in Acute Exacerbations in Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Evaluate Biomarkers in Chronic Obstructive Pulmonary Disease
Status: Terminated | Type: Observational
Why Stopped: Study was completed with 69 subjects enrolled due to difficult enrolment and adequate biomarker data was avaible with 69 subjects in the study.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MI-CP221
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Symptom, physiological data, blood, and sputum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 2: Subjects who are recruited on admission to hospital for AECOPD.
- Cohort 1: Subjects with COPD who are stable, but at risk of presenting with an AECOPD.

SUMMARY:
The primary objective of this study is to identify biomarkers that can be used for evaluation of efficacy in subjects presenting with AECOPD

DETAILED DESCRIPTION:
Identify biomarkers that can be used for evaluation of efficacy in subjects presenting with AECOPD by evaluating longitudinal changes and the interrelationship of blood and sputum biomarkers with physiological endpoints and symptom measures in stable subjects with COPD likely to experience a future AECOPD, and in subjects during severe AECOPD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years at the time of screening
* Written informed consent and any locally required authorization (eg, HIPAA in the USA, EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
* Cohort 1 only: A primary diagnosis of clinically stable physician-diagnosed COPD upon entry into the study meeting one of the following criteria:
* Subjects who have experienced a severe AECOPD requiring inpatient hospitalization in the previous 12 months
* Subject who had one severe AECOPD requiring ED visits in the past 9 months
* Subjects who are currently on LTOT.
* Cohort 1 only: Stable COPD for 4 weeks prior to screening, as defined by no change in ICS therapy and no use of oral corticosteroids or antibiotics for a respiratory tract infection.
* Cohort 1 only: Forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) < 0.70 or lower limits of normal (LLN).
* Cohort 1 only: FEV1 < 60% predicted normal value.
* Cohort 2 only: A primary diagnosis of physician-diagnosed AECOPD requiring admission to the hospital.
* Current smoker or ex-smoker with a tobacco history of ≥ 10 pack-years (one pack year = 20 cigarettes smoked per day for 1 year).
* Ability and willingness to complete the appropriate follow-up period of time as required by the protocol.
* Able to read and write and use the electronic devices (English or Spanish version).

Exclusion Criteria:

* Participation (defined as administration of at least one dose of investigational product) in another clinical study, the last follow-up visit of which is within 12 weeks (for a small molecule drug) and (6 months for a large molecule drug) of entry into this study.
* Any condition that, in the opinion of the investigator would interfere with interpretation of subject safety or study results.
* Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals.
* The presence of another chronic pulmonary or systemic disease, which in the opinion of the investigator or medical monitor might affect the analysis of the data (eg, idiopathic pulmonary fibrosis, sarcoidosis, active cancer or autoimmune disease).
* History of immunodeficiency.
* Current alcohol or drug abuse or a history of unsuccessfully treated alcohol or drug abuse within the past year.
* Cohort 2 only: Diagnosis of an acute disease/condition (eg, congestive heart failure, acute myocardial infarction, pneumonia, or pulmonary embolus) that is the primary reason for the subject's hospitalization.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects in this study will be adult males or females, ≥40 years of age, at increased risk for AECOPD (Cohort 1) or who present with severe AECOPD requiring hospitalization (Cohort 2).
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Identify biomarkers for evaluation of efficacy in subjects presenting with AECOPD | 12 months
  Investigate changes in physiological measures, symptoms, and blood, urine and sputum biomarkers in subjects with stable COPD during AECOPD, and as subjects return to clinical stability.

SECONDARY OUTCOMES:
Hospitalization, treatment and discharge of COPD subjects | 12 months
  Gain an understanding of the reasons subjects with COPD may be hospitalized for their AECOPD and to understand the criteria physicians use for treatment and discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Parker, MD, Study Director — MedImmune LLC
Locations (10):
- United States (9):
  - Research Site, Baltimore, Maryland
  - Research Site, Springfield, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Buffalo, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Houston, Texas
- Research Site, Sainte-Foy, Quebec, Canada